CLINICAL TRIAL: NCT03551639
Title: Application of Real-time PCR Platform for Detection of Vittaforma Corneae Among Patients With Microsporidia Keratitis
Acronym: MK
Status: Withdrawn | Type: Observational
Why Stopped: no patient meet of criteria the trial
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201610011RIND
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Microsporidia Keratitis; Microsporidial Keratoconjunctivitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diagnosis of patients with microsporiosis relies on pathological findings as well as laboratory detection of the causative organism. The conventional laboratory diagnosis of microsporiosis relies on microscopic visualization of the characteristic V. Corneae organisms. We develop a fully automated molecular platform for detection of Vittaforma corneae among patients with microsporidia keratitis.

DETAILED DESCRIPTION:
Clinical infections due to Microsporidium spp. are protean and can be found in humans, insects, and fishes. The most common type of infection is keratitis and mostly is caused by Vittaforma corneae. Diagnosis of patients with microsporiosis relies on pathological findings as well as laboratory detection of the causative organism. The conventional laboratory diagnosis of microsporiosis relies on microscopic visualization of the characteristic V. Corneae organisms. Laboratory tools of identification of V. corneae include Gram staining, Giemsa staining, and modified Ziehl-Neelsen staining of scratching or biopsied specimens of infected cornea. However, the sensitivity of these staining methods is not acceptable due to the variation of specimen quality and quantity, processing, and low load of organisms in the specimens. The BD MAX system (Beckon Dickinson, Diagnostic Systems, Sparks, MD, USA) was introduced in clinical microbiology laboratory of NTUH in 2014 for Pneumocystis jirovecii detection. Till now, no data are available in using this system on V. corneae detection. We develop a fully automated molecular platform for detection of Vittaforma corneae among patients with microsporidia keratitis.

ELIGIBILITY:
Inclusion Criteria:

Patients with suspected microsporidia infection in eye

Exclusion Criteria:

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected microsporidia infection in eye at the National Taiwan University Hospital (NTUH)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Microsporidia spp. analysis | 2016/1/1-2018/12/31
  Corneal scrapings were collected in patients. Gram stain, modiﬁed Kinyoun acid-fast stain, polymerase chain reaction (PCR) and gene analysis of the microsporidian 16S ribosomal RNA (rRNA) were examined for detection of Microsporidia spp.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chun Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan